CLINICAL TRIAL: NCT01136564
Title: Reno- and Vascular Protective Effect of a Low-calcemic Vitamin-D-analogue (Paricalcitol) in Stage III-IV Chronic Kidney Disease
Brief Title: Reno- and Vascular Protective Effect of a Vitamin-D-analogue in Moderate to Severe Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, Professor, MD, MSci, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBP-TL-2010; 2009-017619-14 (EudraCT Number)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Kidney Disease
Keywords: paricalcitol; vitamin d; kidney disease; renin; proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Proteinuria | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol (Active Comparator)
  Interventions: Drug: Zemplar
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zemplar — 2 capsules of 1 microgram daily
  Arms: Paricalcitol
Drug: Placebo — 2 capsules daily
  Arms: Placebo

SUMMARY:
Recently it has been documented that vitamin D has important functions in the human body that are unrelated to its primary effects in calcium homeostasis and bone mineralization. In clinical studies, paricalcitol - a low-calcemic vitamin D analogue - has been shown to decrease proteinuria, a marker of disease progression and cardiovascular risk in patients with chronic kidney disease (CKD). The purpose of this study is to investigate the effect of a paricalcitol on renal and cardiovascular variables in patients with moderate to severe CKD.

ELIGIBILITY:
Inclusion Criteria:

* Kidney disease corresponding to eGFR: 15-59 ml/min
* Albuminuria > 30 mg/l

Exclusion Criteria:

* Total parathyroidectomy
* Diabetes Mellitus
* Cancer
* Illicit drug or alcohol abuse
* Pregnancy og nursing
* Ongoing NSAID or corticosteroid treatment
* b-hemoglobin < 6 mmol/l
* p-albumin < 25 mmol/l
* Clinically significant hypercalcemia
* Office blood pressure > 170/105 mmHg that despite antihypertensive treatment still is > 170/105 mmHg when using home blood pressure measurements or 24-hour ambulatory blood pressure measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
plasma renin concentration | 6 weeks

SECONDARY OUTCOMES:
Urinary albumin excretion | 6 weeks
GFR | 6 weeks
Fractional excretion of sodium | 6 weeks
Urinary excretion of aquaporin-2 | 6 weeks
Urinary excretion of ENaC-beta | 6 weeks
Urinary excretion of NCC | 6 weeks
Plasma concentration of aldosterone | 6 weeks
Plasma concentration of angiotensin-II | 6 weeks
Plasma concentration of ADH | 6 weeks
Plasma concentration of atrial natriuretic peptide | 6 weeks
Plasma concentration of brain natriuretic peptide | 6 weeks
Plasma concentration of endothelin | 6 weeks
24-hr ambulatory blood pressure | 6 weeks
Central blood pressure | 6 weeks
Pulse wave velocity | 6 weeks
augmentation index | 6 weeks
Plasma concentration of ionized calcium | 6 weeks
Plasma concentration of phosphate | 6 weeks
Plasma concentration of alkaline phosphatase | 6 weeks
Plasma concentration of Parathyroid hormon | 6 weeks
Plasma concentration of 25-hydroxy-vitamin D | 6 weeks
Plasma concentration of ultrasensitive CRP | 6 weeks
Plasma concentration of TNF-alpha | 6 weeks
Plasma concentration of TGF-beta | 6 weeks
Urinary excretion of calcium | 6 weeks
Plasma concentration of ADMA | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Prof, MSci, Principal Investigator — Department of Medical Research
Locations (1):
- Department of Medical Research, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Larsen T, Mose FH, Bech JN, Pedersen EB. Effect of paricalcitol on renin and albuminuria in non-diabetic stage III-IV chronic kidney disease: a randomized placebo-controlled trial. BMC Nephrol. 2013 Jul 26;14:163. doi: 10.1186/1471-2369-14-163. PMID 23889806